CLINICAL TRIAL: NCT03472248
Title: Smartphone Delivered Acceptance and Commitment Therapy for Adolescents With Longstanding Pain - a Pilot Study
Brief Title: Smartphone Delivered Acceptance and Commitment Therapy for Adolescents With Longstanding Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Rikard Wicksell, Associate Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017/1676-31/2
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Chronic Pain
Keywords: Adolescents; Acceptance and Commitment Therapy; Smartphone
MeSH Terms: conditions — Chronic Pain | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acceptance and Commitment Therapy (Experimental): Eight weeks of smartphone delivered Acceptance and Commitment Therapy for the adolescent and eight weeks of internet delivered parental support to one or two parents of the adolescent.
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Eight weeks of smartphone delivered Acceptance and Commitment Therapy for the adolescent and eight weeks of internet delivered parental support to one or two parents of the adolescent.

SUMMARY:
Intervention study with uncontrolled design investigating the effects of smartphone delivered Acceptance and Commitment Therapy for longstanding pain in adolescents. Primary outcome is pain interference. Internet-based parental support will be offered to the adolescents' caregivers.

ELIGIBILITY:
Inclusion Criteria:

* pain duration of ≥ 3 months;
* the pain condition has been examined by a medical doctor
* able to communicate in Swedish
* access to a smartphone and internet connection on a daily basis
* stable medication use since 2 months time, with no planned changes

Exclusion Criteria:

* previous ACT or CBT treatment during the past 6 months
* severe psychiatric co-morbidity (e.g. psychosis or high risk of suicide) as assessed by the psychologist in a semi-structured interview

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2019-09-19 (Actual)

PRIMARY OUTCOMES:
Pain Interference Index (PII) | Pre-treatment, weekly for eight weeks (during treatment), after 8 weeks (i.e. post-treatment), 8 weeks and 4 months after treatment is completed (i.e. 4 months follow-up), 8 weeks and 1 year after treatment (i.e. 1 year follow-up)
  Change in pain interference on the adolescent daily activities. Items are rated on a 7-point Likert scale, and the total score is the mean of the completed items. Higher scores indicate more interference.

SECONDARY OUTCOMES:
Pediatric Quality of Life Inventory (PedsQL) | Pre-treatment, after 8 weeks (i.e. post-treatment), 8 weeks and 4 months after treatment is completed (i.e. 4 months follow-up), 8 weeks and 1 year after treatment (i.e. 1 year follow-up)
  Change in quality of life for the adolescent. This questionnaire is composed of four subscales: Physical functioning (8 items), Emotional functioning (5 items), Social functioning (5 items), and School functioning (5 items). Each item has a scoring between 0 and 4, where a higher score indicate a better health-related quality of life. The subscales are summed together to a total score.
Center for Epidemiological Studies Depression Scale for Children (CES-DC) | Pre-treatment, after 8 weeks (i.e. post-treatment), 8 weeks and 4 months after treatment is completed (i.e. 4 months follow-up), 8 weeks and 1 year after treatment (i.e. 1 year follow-up)
  Change in depressive symptoms for the adolescent. Scores on the CES-DC are summed to a total score, ranging from 0 to 60, in which higher scores suggest a greater presence of depressive symptoms.
Insomnia Severity Index (ISI) | Pre-treatment, after 8 weeks (i.e. post-treatment), 8 weeks and 4 months after treatment is completed (i.e. 4 months follow-up), 8 weeks and 1 year after treatment (i.e. 1 year follow-up).
  Change in insomnia severity for the adolescent. Scores on the seven items are summed into a total score, ranging from 0 to 28, where higher scores indicate greater severity of insomnia.
Psychological Inflexibility in Pain Scale (PIPS) | Pre-treatment, weekly for eight weeks (during treatment), after 8 weeks (i.e. post-treatment), 8 weeks and 4 months after treatment is completed (i.e. 4 months follow-up), 8 weeks and 1 year after treatment (i.e. 1 year follow-up)
  Change in psychological flexibility for the adolescent. PIPS is composed on two subscales: Avoidance (8 items) and Defusion (4 items). Each item has a scoring ranging between 0 and 6. Scores are summed into subscales and into a total scale. Higher scores indicate higher degree of psychological inflexibility.

OTHER OUTCOMES:
Pain Reactivity Scale - Parent (PRS-P) | Pre-treatment, after 8 weeks (i.e. post-treatment), 8 weeks and 4 months after treatment is completed (i.e. 4 months follow-up), 8 weeks and 1 year after treatment (i.e. 1 year follow-up)
  Change in pain reactivity for the parent in relation to the child's pain. Each of the five items of the PRS-P is rated on a scale from 0 to 6, and summed together, with a maximum total score of 30. Higher scores indicate more pain reactivity.
Parent Psychological Flexibility Questionnaire (PPFQ) | Pre-treatment, after 8 weeks (i.e. post-treatment), 8 weeks and 4 months after treatment is completed (i.e. 4 months follow-up), 8 weeks and 1 year after treatment (i.e. 1 year follow-up)
  Change in psychological flexibility for the parent. A ten item questionnaire, with item scoring between 0 and 6. The PPFQ is summed into three subscales: Emotional acceptance (4 items), Values-based action (3 items), and Pain willingness (3 items). The subscales are also summed to a total score, where higher scores indicate more flexibility.
Patient Health Questionnaire (PHQ-9) | Pre-treatment, after 8 weeks (i.e. post-treatment), 8 weeks and 4 months after treatment is completed (i.e. 4 months follow-up), 8 weeks and 1 year after treatment (i.e. 1 year follow-up)
  Change in depressive symptoms for the parent. PHQ-9 is a nine item inventory summed into a total scale, with scores ranging from 0 to 27. Higher scores indicate more depressive symptoms.
Generalized Anxiety Disorder (GAD-7) | Pre-treatment, after 8 weeks (i.e. post-treatment), 8 weeks and 4 months after treatment is completed (i.e. 4 months follow-up), 8 weeks and 1 year after treatment (i.e. 1 year follow-up)
  Change in anxiety symptoms for the parent. GAD-7 is a seven item inventory summed into a total scale, with scores ranging from 0 to 21. Higher scores indicate more anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Rikard Wicksell, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No